CLINICAL TRIAL: NCT00679250
Title: A Placebo Controlled Trial to Evaluate The Effects of Levocetirizine on Nasal Allergen Challenge And Adenosine Monophosphate Challenge In Patients With Intermittent and Persistent Allergic Rhinitis
Brief Title: To Evaluate Adenosine Monophosphate and Allergen Challenge in Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brian J Lipworth (Other)
Responsible Party: Sponsor-Investigator, Brian J Lipworth, Professor (Clinical) Airway allergy and COPD, University of Dundee
Organization: University of Dundee (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: GRAY09; 2004-000683-27
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Allergic Rhinitis
Keywords: allergic rhinitis; levocetirizine; nasal provocation testing; nasal allergen challenge; nasal adenosine monophosphate challenge
MeSH Terms: conditions — Rhinitis, Allergic | interventions — levocetirizine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levocetirizine (Experimental): Active drug
  Interventions: Drug: levocetirizine
- placebo (Placebo Comparator): placebo to levocetirizine
  Interventions: Drug: placebo to levocetirizine

INTERVENTIONS:
Drug: levocetirizine — 5 mg once nightly before visit
  Arms: Levocetirizine
Drug: placebo to levocetirizine — 1 tablet once nightly before visit
  Arms: placebo

SUMMARY:
Allergic rhinitis is a common condition characterize by inflammation of the upper airways. Third generation antihistamines have been demonstrated effective in the treatment of this condition. Allergen challenge can be use to assess the effects of drugs in allergic rhinitis, adenosine monophosphate may also be used as a means to investigate these effects but as yet its effects have yet to be compared to allergen challenge. We intend to compare the effects of levocetirizine at a single dose of 5mg on allergen and AMP challenge compared to placebo in a double blind cross-over study. The study will include 20 patients with allergic rhinitis. Each patient will have allergen and AMP challenge on placebo and active treatment. The primary outcome variable will be the change in concentration of AMP/Allergen required to produce a 20% drop in nasal flow as manifest by peak nasal inspiratory flow. A 1 doubling dose change in concentration of challenge medium to cause a 20% drop in nasal flow will be deemed significant. We will also measure time to recovery after both challenges. AMP challenge is a safe alternative to allergen challenge and does not have the risk of anaphylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 16-75
* Patients with persistent rhinitis must be skin prick positive to house dust mite with perennial symptoms
* Patients with seasonal rhinitis should be skin prick positive to grass/tree pollen with seasonal symptoms
* Concomitant asthma is permitted in those with rhinitis if FEV1 >60%
* No recent exacerbations of asthma or chest infections if asthmatic
* Able to perform all of the techniques necessary to carry out challenge testing
* Must be compliant to study medication
* Must give informed consent

Exclusion Criteria:

* Male or female outwith the above age range
* Negative skin prick testing
* Patients with concomitant asthma with FEV1 less than 60% predicted
* Patients with asthma with recent chest infection or exacerbation
* Pregnant females, those at risk of becoming pregnant or breast feeding. Females must be on adequate contraception for the whole study period

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-11; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Provocative concentration of AMP or Allergen required to cause a 20% drop in Peak Nasal Inspiratory Flow. | 1 hour

SECONDARY OUTCOMES:
Recovery Time Profile after nasal AMP and Allergen challenge | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Arun Nair, MRCP, Principal Investigator — University of Dundee
Locations (2):
- United Kingdom (2):
  - Ninewells Hospital and Medical School (Tayside NHS Trust, University of Dundee), Dundee, Angus
  - Perth Royal Infirmary, Perth, Perthshire

REFERENCES:
- [Background] Togias A. Rhinitis and asthma: evidence for respiratory system integration. J Allergy Clin Immunol. 2003 Jun;111(6):1171-83; quiz 1184. doi: 10.1067/mai.2003.1592. PMID 12789212
- [Background] Bousquet J, Van Cauwenberge P, Khaltaev N; Aria Workshop Group; World Health Organization. Allergic rhinitis and its impact on asthma. J Allergy Clin Immunol. 2001 Nov;108(5 Suppl):S147-334. doi: 10.1067/mai.2001.118891. No abstract available. PMID 11707753
- [Background] Clough GF, Boutsiouki P, Church MK. Comparison of the effects of levocetirizine and loratadine on histamine-induced wheal, flare, and itch in human skin. Allergy. 2001 Oct;56(10):985-8. doi: 10.1034/j.1398-9995.2001.00204.x. PMID 11576078
- [Background] Wang DY, Hanotte F, De Vos C, Clement P. Effect of cetirizine, levocetirizine, and dextrocetirizine on histamine-induced nasal response in healthy adult volunteers. Allergy. 2001 Apr;56(4):339-43. doi: 10.1034/j.1398-9995.2001.00775.x. PMID 11284803
- [Background] Lee DK, Gray RD, Wilson AM, Robb FM, Soutar PC, Lipworth BJ. Single and short-term dosing effects of levocetirizine on adenosine monophosphate bronchoprovocation in atopic asthma. Br J Clin Pharmacol. 2004 Jul;58(1):34-9. doi: 10.1111/j.1365-2125.2004.02110.x. PMID 15206990
- [Background] Terada N, Hamano N, Kim WJ, Hirai K, Nakajima T, Yamada H, Kawasaki H, Yamashita T, Kishi H, Nomura T, Numata T, Yoshie O, Konno A. The kinetics of allergen-induced eotaxin level in nasal lavage fluid: its key role in eosinophil recruitment in nasal mucosa. Am J Respir Crit Care Med. 2001 Aug 15;164(4):575-9. doi: 10.1164/ajrccm.164.4.2009046. PMID 11520718
- [Background] Wilson AM, Sims EJ, Orr LC, Robb F, Lipworth BJ. An evaluation of short-term corticosteroid response in perennial allergic rhinitis using histamine and adenosine monophosphate nasal challenge. Br J Clin Pharmacol. 2003 Apr;55(4):354-9. doi: 10.1046/j.1365-2125.2003.01776.x. PMID 12680883
- [Result] Vaidyanathan S, Nair A, Barnes ML, Meldrum K, Lipworth BJ. Effect of levocetirizine on nasal provocation testing with adenosine monophosphate compared with allergen challenge in allergic rhinitis. Clin Exp Allergy. 2009 Mar;39(3):409-16. doi: 10.1111/j.1365-2222.2008.03166.x. PMID 19187327